

## **Participant Consent Form**

## Project: Digital Lens Research

Please read the following statements and initial each box to confirm your agreement:

| I confirm that I have read the participant information sheet dated (20/04/2022) for the above study. I have had the opportunity to consider the information, | |
|---|---|
| ask questions and have had these answered satisfactorily. | |
| I am aware that my responses will be anonymised and an anonymous pooled | |
| data set will be created and will be used within a project report and may | |
| feature in other academic outputs such as, conference presentations and | |
| professional journal publications. | |
| I am aware that my participation is voluntary, and I have the right to withdraw | |
| before the final data collection visit takes place. However, information that | |
| has been submitted before withdrawal may already be anonymised and it will | |
| not be possible to remove it. | |
| I am aware I do not have to provide any reason for withdrawing from the | |
| study. | |
| I understand that I will have to attend five (5) separate data collections | |
| sessions over a 16-week period, if I take part in the above study | |
| I agree to take part in the above study. | |
| If you have used and wedenates of this services forms and some to moutising | 4- : 41-:- |
| If you have read and understood this consent form and agree to participa | te in this |
| research, please sign below, | |
| Name of Participant: | |
| Name of Fartiopant. | |
| Signed: Date: | |
| Name of Researcher: | |
| Name of Nessalonon | |
| Signed: Date: | |